CLINICAL TRIAL: NCT00600431
Title: Melanocytic-Nevi-Counts During Chemotherapy of Children With Malignancies.
Brief Title: Melanocytic Nevi in Children Under Chemotherapy
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Binder Barbara, MD, Department of Dermatology and Department of Pediatric Oncology, MU Graz
Other Study IDs: 001
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Nevus, Pigmented
Keywords: nevus count; children; chemotherapy
MeSH Terms: conditions — Nevus, Pigmented

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Study group: 16 children under 18 years undergoing systemic chemotherapy
- 2: Control group: 16 age and sex matched healthy children under 18 years

SUMMARY:
Changes in nevus count in 16 children (8m, 8f) aged between 2 and 17 years (median:8 years) suffering from different malignancies were examined every three months during a one-year period after starting chemotherapy. An age and sex matched control group underwent the same skin examinations.At the start of our study, the range of number of nevi in the chemotherapy group was 0-133, in the control group 2-199.

DETAILED DESCRIPTION:
Objectives:

Patients given chemotherapy because of different malignancies have an increased susceptibility to cutaneous tumours and infection and a change of number of nevi during treatment is discussed. We investigated wether total nevi count changes in children undergoing chemotherapy. Therefore 16 (8m, 8f) children suffering from leukaemia (11), lymphoma (2), adenosarcoma of the kidney (1), Ewing´s sarcoma (1) and neuroblastoma (1) aged between 2 and 17 years (median:8 years), under chemotherapy at the pediatric department of oncology, were examined at the beginning and 9-12 months after starting chemotherapy. As control group age and sex matched children of the local population were used.

Materials and Methods:

At the beginning of chemotherapy the nevi were counted on the total body. All nevi were larger in diameter than 1mm and as melanocytic lesion identifiable. Clinical and dermoscopic photographs were taken of every nevus. If the patient had more than 50 nevi, only nevi on the face, right arm, upper back and the buttocks were documented. Reassessment was repeated every 3 month.

Conclusion:

In our patients under chemotherapy during one year the development of new nevi is similar to sex and age matched children of the general population. During this short period development of nevi seems not to be influenced by chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient and/or parents willing to participate in the study
* Age under 18

Study Group Only:

* Patient suffering from a malignancy requiring systemic chemotherapy

Exclusion Criteria:

* Patient and/or parents who decline to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study group: children suffering from malignancies requiring chemotherapy were recruited consecutively at the department of pediatric oncology
  Control group: children were recruited consecutively at our department for pigmented skin lesions at the department of dermatology
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
total body nevus count | Every three months during a one year period

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Binder, MD, Study Chair — Department of Dermatology, Medical University of Graz, Austria
Locations (1):
- Department of Dermatology, Medical University of Graz, Graz, Austria